CLINICAL TRIAL: NCT01381640
Title: A Single Dose Pharmacoscintigraphic Study Investigating the Differences in Gastrointestinal Behavior and Paracetamol Absorption Between Sustained Release Formula and Standard Release Formula
Brief Title: A Study to Compare Two Paracetamol Tablets
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was cancelled prior to enrolling any subjects.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A4040689
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Subjects
Keywords: paracetamol; healthy volunteer; pharmacoscintography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed paracetamol (Active Comparator): Marketed formulation
  Interventions: Drug: Marketed paracetamol
- Experimental paracetamol formulation (Experimental): Experimental formulation
  Interventions: Drug: Experimental paracetamol formulation

INTERVENTIONS:
Drug: Marketed paracetamol — marketed formulation
  Arms: Marketed paracetamol
Drug: Experimental paracetamol formulation — Experimental formulation
  Arms: Experimental paracetamol formulation

SUMMARY:
This is a single dose pharmacoscintigraphic study investigating the differences in paracetamol absorption between two formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who are in good general health
* Have not exceeded the limits of total radiation exposure (5mSv) allowed in any 12 month period

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Time of onset and completion of disintegration based on release of radiolabeled markers in a fed condition | Baseline to 12 hours post dosing

SECONDARY OUTCOMES:
To assess the gastrointestinal transit by qualitative scintigraphic analysis | Baseline to 12 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - BIO-IMAGES Research Ltd., Glasgow, Scotland
  - Bio-Images, Glasgow, Scotland